CLINICAL TRIAL: NCT05456698
Title: Efficacy and Safety of Inotuzumab Ozogamicin in Treating Adult Patients With Ph Negative ALL With Minimal Residual Disease Positive After Induction Chemotherapy: A Phase 2, Open-label, Single-arm, Single-center Trial
Brief Title: Efficacy and Safety of Inotuzumab Ozogamicin in Treating Adult Patients With Ph Negative ALL With Minimal Residual Disease Positive After Induction Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022011
Record Dates: First submitted 2022-03-29; First posted 2022-07-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inotuzumab Ozogamicin (Experimental): Each subject will be treated with Inotuzumab Ozogamicin
  Interventions: Drug: Inotuzumab ozogamicin

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — Patients who achieved CR/CRi had their InO dose at 1.5mg/m2 per cycle (28days/cycle), with 0.5mg/m2 administered on days 1, 8, and 15.
  Patients received treatment for up to two cycles in the absence of disease progression or unacceptable toxicity.
  Other Names: CMC-544

SUMMARY:
A single-center, single-arm, open-label, interventional, phase II clinical trial to evaluate the efficacy and safety of InO in B-ALL achieved CR/CRi after 1L induction chemotherapy with positive minimal residual disease.

ELIGIBILITY:
Inclusion Criteria:

1. New diagnosed B-ALL in hematologic complete remission (CR) after 1L induction chemotherapy with MRD positive. Molecular disease or MRD is defined by a value of at least of 10-4 (0.01%) by multicolor flow cytometry.
2. Age ≥18 years
3. ECOG PS score: 0 to 2
4. Functions of the main organs are normal, if the following criteria are met:

   1. Total bilirubin (BIL) ≤ 1.5 × upper limit of normal (ULN)
   2. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × ULN
   3. Serum creatinine ≤ 1.5 × ULN
   4. Creatinine clearance ≥ 30 ml/min
5. No active or co-existing malignancy with a life expectancy of less than 12 months
6. Patients are voluntarily enrolled into the study and have good compliance, and the Informed Consent Form (ICF) needs to be signed.

Exclusion Criteria:

1. Mixed lineage leukemia
2. Clinically significant liver disease such as history of veno-occlusive disease (VOD)/ sinusoidal obstruction syndrome (SOS)
3. Patients with severe and / or uncontrolled diseases, such as:

   1. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmias; uncontrolled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)
   2. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis
   3. Known to be human immunodeficiency virus positive (HIV+)
   4. Active and uncontrolled disease/infection as judged by the treating physician
   5. Active central nervous system (CNS) or extramedullary disease
   6. Patients who have other malignant tumors at the same time; patients who are evaluated by the investigator to have concomitant diseases that seriously endanger the safety of the patients or affect the patients to complete the study
4. Pregnant or nursing women
5. Unable or unwilling to sign the consent form
6. Monoclonal antibodies therapy within 2 weeks before study entry
7. Radiotherapy or cancer chemotherapy (except for induction chemo) or any investigational drug within 2 weeks before study entry
8. Patients who have severe allergies (≥ grade 3) to active ingredients and any excipients of InO
9. Patients in other situations who are evaluated by the investigator to be ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2030-11-05 (Estimated)

PRIMARY OUTCOMES:
MRD negativity rate within the first treatment cycle | At the end of Cycle 1 (each cycle is 28 days)
  MRD negativity is defined as no presence of small numbers of leukemic cells detected by the flow cytometry after remission

SECONDARY OUTCOMES:
Complete MRD response rates | At the end of Cycle 1 and Cycle 2, respectively (each cycle is 28 days)
  Complete MRD response is defined as no presence of small numbers of leukemic cells detected by the flow cytometry after remission
Duration of MRD negativity rate | From enrollment to the end of Cycle 1 or Cycle 2, which achieves MRD negative first (each cycle is 28 days)
  The duration of MRD response was analyzed as the time from onset of MRD negativity until MRD or hematological relapse or date of last confirmation of negative MRD status.
MRD level variation from baseline to post cycle 1, cycle 2 in patients with detectable MRD, respectively | From enrollment to the end of Cycle 1 and Cycle 2, respectively (each cycle is 28 days)
  The variation of MRD level from baseline to post cycle 1, cycle 2, respectively
Relapse-free Survival (RFS) | Up to 5 years from enrollment
  RFS is defined as the time from the date of CR until the date of relapse or death
Overall Survival (OS) | Up to 5 years from enrollment
  OS is defined as the time from enrollment to date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No